CLINICAL TRIAL: NCT04323033
Title: Prospective, Randomized Clinical Trial Evaluating Safety and Efficacy of Cobalt-chromium Sirolimus Eluting Stent (PERS) by Balton Versus Cobalt-chromium Stent (Neptune C), to Maintain Patency of Iliac Arteries in Patients Undergoing Peripheral Angioplasty
Brief Title: Safety and Efficacy of Peripheral, Cobalt-chromium Sirolimus Eluting Stent (PERS) Versus Cobalt-chromium Stent (Neptune C)
Acronym: PERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERS
Record Dates: First submitted 2019-10-16; First posted 2020-03-26 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERS stent (Experimental): 20 Patients will receive PERS stent
  Interventions: Device: PERS stent
- NEPTUN C stent (Active Comparator): 20 Patients will receive NEPTUN C stent
  Interventions: Device: NEPTUN C stent

INTERVENTIONS:
Device: PERS stent — PERS® is a cobalt-chromium stent, made of cobalt-chromium alloy with drug (Sirolimus) and biodegradable polymer controlling drug elution.
  The length of the stent is selected to cover the treated lesion with a margin of 5 mm proximal and distal, while the diameter of the stent will be selected based on the QVA measurement (balloon to vessel ratio 1:1).
  Arms: PERS stent
Device: NEPTUN C stent — Neptun C is balloon-expanding cobalt-chromium stent.
  Arms: NEPTUN C stent

SUMMARY:
The aim of this study is to assess the safety and efficacy of PAD treatment by revascularization with new cobalt-chromium sirolimus stent implantation, which is expandable on balloon PERS (CoCr SES) compared to cobalt-chromium balloon-expandable (Neptun C) stent (CoCr BMS) in patients with symptomatic iliac arteries disease requiring revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. De novo lesion or restenosis without previously implanted stent, in a common or external iliac artery with a reference diameter of 5 to 12 mm, length up to 10 cm and stenosis ≥ 50% and ≤ 99% (in quantitative assessment by peripheral angiography), which may be treated with one stent or total occlusion of vessels up to 50 mm long.
2. Ability to cross the lesion with guidewire (assessed during diagnostic angiography).
3. ABI ankle-brachial index <0.9.
4. Signs of lower limb ischemia based on the Rutherford scale in the range from 2 to 4.
5. Age ≥ 18 years.
6. Patient signed informed consent form.

Exclusion Criteria:

1. Life expectancy less than two years.
2. Chronic kidney disease in stage III-V.
3. Lesion in the previously implanted by-pass.
4. Target lesion is a chronic total occlusion of significant length, not eligible for percutaneous revascularization.
5. Acute lower limb ischemia.
6. Stenosis (> 50%) or occlusion proximally to the lesion being treated.
7. Angiographically confirmed thrombus in the lesion to be treated.
8. Treatment requires an atherectomy to deliver stent to treated lesion.
9. Known allergy or hypersensitivity to clopidogrel.
10. Hemorrhagic stroke in the last three months.
11. Contraindications for acetylsalicylic acid (hypersensitivity, hemorrhagic diathesis).
12. Pregnancy or women of childbearing potential not using effective contraception.
13. Active inflammation at the planned access site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of MAE | 12 months FU
  Occurrence of major adverse event (MAE) in 12 months follow up, defined as death related to stent implantation of procedure, amputation above metatarsus in treated limb due to vascular complication or/and reintervention in treated lesion (TLR).

SECONDARY OUTCOMES:
Vessel patency | 30 days, 6 months and 12 months FU
  Vessel patency 30 days, 6 and 12 months after the initial procedure assessed by Dupplex Doppler
Success of implanting the device | Directly after implantation, at the end of endovascular index procedure
  Success of implanting the device, defined as residual stenosis ≤30% in angiographic assessment.
Procedural success | Up to 7 days after procedure
  Procedural success, defined as residual stenosis ≤30% in angiographic assessment and lack of procedurę related SAE.
Clinical success | During follow-up visits: 30 days, 6 months and 12 months
  Clinical success, defined as improvement in Rutherford classification for at least 1 point.
ABI (ankle-brachial index) change | 30 days and 12 months FU
  ABI (ankle-brachial index) change after 30 days and 12 months
Mortality rate | 30 days, 6 months and 12 months FU
  Mortality rate after 30 days, 6 months and 12 months (cardiovascular deaths)
Artery patency in Duplex Doppler USG: Maximum velocity flow | 30 days, 6 months and 12 months FU
  Maximum velocity flow assessed by Dupplex Doppler
Artery patency in Duplex Doppler USG: % of diameter stenosis | 30 days, 6 months and 12 months FU
  % of diameter stenosis (DS in target lesion) assessed by Dupplex Doppler

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Małopolskie Centrum Sercowo-Naczyniowe PAKS American Heart of Poland S.A., Chrzanów
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin
  - Szpital Eskulap Centrum Leczenia Chorób Serca i Naczyń, Osielsko

IPD SHARING:
Plan to Share IPD: No